CLINICAL TRIAL: NCT00217191
Title: Ibuprofen and Renal Function in Premature Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maternite Regionale Universitaire (Other)
Collaborators: Central Hospital, Nancy, France (Other); Ministere de la Sante et de la Protection Sociale, France (Unknown)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MRAP040833; PHRC2004:17-06
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Premature Infants; Patent Ductus Arteriosus
Keywords: Premature Infants; Patent ductus arteriosus; Renal function; Ibuprofen
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent | interventions — Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen

SUMMARY:
Purpose of the study:

1. To evaluate renal function maturation within the first month of life in very premature infants.
2. To determine whether a treatment with Ibuprofen for patent ductus arteriosus would alter renal function maturation at short term and up to 28 days of life.

DETAILED DESCRIPTION:
Ibuprofen has improved the prognosis of infants with Patent Ductus Arteriosus. Several studies showed that Ibuprofen has significantly less side effects than Indomethacin that was used for this indication. However, experimental studies and few clinical observations suggested that side effects on renal function could occur in very premature infants.

Purpose of the study:

1. To evaluate renal function maturation within the first month of life in very premature infants.
2. To determine whether a treatment with Ibuprofen for patent ductus arteriosus would alter renal function maturation at short term and up to 28 days of life.

Population:

At least 120 infants 27 to 31 weeks gestation will be studied. That number will allow to demonstrate a 30% difference in creatinine clearance on day 7 postnatally. Careful recording of mother and child history, and associated therapies prone to alter renal function should allow to improve the use of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age = 27 to 31 weeks
* Postnatal age < 48 hours
* Parental Consent Obtained

Exclusion Criteria:

* Renal malformation
* Urinary tract infection
* Renal Failure
* Pulmonary Hypertension at echocardiography

Ages: 0 Years to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 2004-09; Study Completion 2006-09

PRIMARY OUTCOMES:
Creatinine Clearance on day seven postnatally

SECONDARY OUTCOMES:
Rate of ductus closure after treatment
Mortality
Rate of necrotizing enterocolitis
Rate and severity of Intraventricular Hemorrhage
Renal function maturation over 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel HASCOET, MD, Study Director — University of Nancy, France
Locations (3):
- France (3):
  - CHU, Dijon
  - AP-HM (Néonatologie), Marseille
  - Maternite Regionale Universitaire, Nancy

REFERENCES:
- [Background] Gournay V, Roze JC, Kuster A, Daoud P, Cambonie G, Hascoet JM, Chamboux C, Blanc T, Fichtner C, Savagner C, Gouyon JB, Flurin V, Thiriez G. Prophylactic ibuprofen versus placebo in very premature infants: a randomised, double-blind, placebo-controlled trial. Lancet. 2004 Nov 27-Dec 3;364(9449):1939-44. doi: 10.1016/S0140-6736(04)17476-X. PMID 15567009
- [Derived] Desandes R, Jellimann JM, Rouabah M, Haddad F, Desandes E, Boubred F, Semama DS, Vieux R, Hascoet JM. Echocardiography as a guide for patent ductus arteriosus ibuprofen treatment and efficacy prediction. Pediatr Crit Care Med. 2012 May;13(3):324-7. doi: 10.1097/PCC.0b013e31822882b5. PMID 21760564
- [Derived] Vieux R, Hascoet JM, Merdariu D, Fresson J, Guillemin F. Glomerular filtration rate reference values in very preterm infants. Pediatrics. 2010 May;125(5):e1186-92. doi: 10.1542/peds.2009-1426. Epub 2010 Apr 5. PMID 20368313
- [Derived] Vieux R, Desandes R, Boubred F, Semama D, Guillemin F, Buchweiller MC, Fresson J, Hascoet JM. Ibuprofen in very preterm infants impairs renal function for the first month of life. Pediatr Nephrol. 2010 Feb;25(2):267-74. doi: 10.1007/s00467-009-1349-9. Epub 2009 Nov 10. PMID 19902266